CLINICAL TRIAL: NCT04027608
Title: Sensitization of the Reinforcing Value of Food as a Predictor of Weight Change in Adolescents
Brief Title: Study of Nutrition and Activity in Kids
Acronym: SNAK
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennifer Temple, Associate Professor, State University of New York at Buffalo
Other Study IDs: STUDY00000042; R01DK106265 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Obesity, Adolescent; Adolescent Behavior
Keywords: adolescent; obesity; relative reinforcing value; physical activity; weight change
MeSH Terms: conditions — Pediatric Obesity; Adolescent Behavior; Obesity; Motor Activity; Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reinforcing value of HED and LED foods in response to snack food monotony — Each child will be asked to eat two different snack foods over the course of two weeks each. The RRV of that food (vs alternative reinforcer) will be tested and baseline and post exposure. Increases in RRv for food after monotony will be considered sensitization to that food. All children will be followed to observe weight change over time for 2 years each.

SUMMARY:
While a substantial body of research suggests that RRV is related to obesity, there is very little research on factors that contribute to the RRV of food, particularly how patterns of eating can increase or decrease the motivation to eat specific foods. Previous work has demonstrated that a subset of individuals with obesity show increases in RRV of food after repeated consumption of large portions of high energy density (HED) snack foods, which has been conceptualized as sensitization. Preliminary data suggest that sensitization of the RRV of HED food is a predictor of weight gain over time. However, more work needs to be done to address this relationship using a planned, prospective study design, using adolescent research subjects, and examining potential moderators of this relationship.

The purpose of this study is to identify risk and protective factors to excess zBMI change in adolescents over time. Aim 1 was to measure the relative reinforcing value (RRV) of a preferred HED and low energy density (LED) snack food before and after 2-weeks of daily exposure. Aim 2 was to assess the RRV of exercise and sedentary activity. Hypotheses include 1) sensitization to HED food will be associated with greater zBMI at the time of testing as well as greater zBMI change over time 2) sensitization to LED food will be associated with lower zBMI at the time of testing in adolescents and less zBMI change over time. 3) Greater RRV of exercise will be protective against zBMI increases over time.

ELIGIBILITY:
Inclusion Criteria:

* between 12-14yoa (male and female)
* zBMI: -1.5 to +2.0 (*determined by Height/weight measurement at Visit 1)
* neutral or higher liking of the study foods
* Willingness to complete 9 study visits over 2 years.

Exclusion Criteria:

* -metabolic or endocrine disorder
* use of medications known to effect appetite (Ritalin, Adderall, Concerta, Wellbutrin, Prednisone, etc)
* Unwilling to complete the study visits
* allergy to study foods
* dislike of study foods (*determined via Preference for Study foods forms at Visit 1)
* parent report that child reads below 4th grade reading level
* parent report that child cannot complete light physical activity without assistance
* No English Speaking parent or legal guardian (therefore cannot provide consent in English nor answer questionnaires for this study) * all other exclusion criteria are assessed from Survey monkey screening in advance of the first appointment vis parental report. At the first appointment the child is directly asses for height, weight, and The linking of study foods.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents living in the Western New York area, aged 12-14 years at the time of enrollment. Flyers were posted in the community within a 30 min drive of UB South Campus. Additionally, flyers were sent to list serves, posted on facebook, and distributed to both private and public schools within a 40 min drive of the university campus.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-28 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balantekin KN, Andrade ALP, Ziegler AM, Temple JL. Restriction and Pressure to Eat Are Associated Cross-Sectionally, But Not Longitudinally, With BMI z-Score in a Longitudinal Cohort Study of Adolescents. Child Obes. 2024 Sep;20(6):386-393. doi: 10.1089/chi.2023.0108. Epub 2023 Nov 15. PMID 37967392
- [Derived] Temple JL, Ziegler AM, Crandall AK, Mansouri T, Hatzinger L, Barich R, Epstein LH. Sensitization of the reinforcing value of high energy density foods is associated with increased zBMI gain in adolescents. Int J Obes (Lond). 2022 Mar;46(3):581-587. doi: 10.1038/s41366-021-01007-w. Epub 2021 Nov 30. PMID 34848836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 201 boys and girls aged 12 - 14 years without obesity recruited using flyers, e-mail and social media, personal referrals, and advertisements distributed in schools in the Buffalo, NY area.
Groups:
- Satiators: Participants who decreased responding for high energy density food after consuming it every day for 2 weeks.
- Sensitizers: Participants who increased responding for high energy density food after consuming it every day for 2 weeks.
Period: Overall Study
Arm/Group | Satiators | Sensitizers
Started | 165 | 36
Completed | 129 | 29
Not Completed | 36 | 7
Not completed — Withdrawal by Subject | 13 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 20 | 4

BASELINE CHARACTERISTICS:
Population: Participants with complete baseline data were included in this analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Satiators | Sensitizers | Total
Number analyzed (Participants) | 165 | 36 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (0.827) | 13.2 (0.845) | 13.3 (0.828)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 16 | 104
  Male | 77 | 20 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaska Native | 1 | 0 | 1
  Race: Asian/Pacific Islander | 3 | 0 | 3
  Race: Black/African American | 20 | 3 | 23
  Race: White or Caucasian | 127 | 33 | 160
  Race: Other/Mixed Race | 14 | 0 | 14
Region of Enrollment [Number; unit: participants]
  United States | 165 | 36 | 201
zBMI [Mean (Standard Deviation); unit: z score] — zBMI was calculated using national standards with '0' being the middle value. A positive zBMI reflects a BMI that is higher than the national average for each sex and age and a negative zBMI reflects a BMI that is lower than the national average for each sex and age.
  z score | 0.38 (1.02) | 0.48 (0.84) | 0.40 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: zBMI Change
Description: BMI z-score change over time. zBMI is a standardized index of body mass index used in children that is standardized to age and sex specific measurements from a national sample. 0 represents the national average. A positive number reflects a body mass index that is higher than the national average and a negative number reflects a body mass index that is lower than the national average.
Time Frame: through study completion, an average of 24 months from baseline.
Population: We began with 165 and 36, but we lost several participants in each group for various reasons which are outlined in an earlier section.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Satiators | Sensitizers
Number analyzed (Participants) | 165 | 36
z-score
  6 months: number analyzed (Participants) | 156 | 35
  6 months | 0.433 (0.073) | 0.55 (0.14)
  15 months: number analyzed (Participants) | 146 | 32
  15 months | 0.376 (0.093) | 0.61 (0.18)
  24 months: number analyzed (Participants) | 129 | 29
  24 months | 0.416 (0.11) | 0.593 (0.25)

ADVERSE EVENTS:
Time Frame: Through study completion up to 24 months.
Description: We used the standard definitions of adverse events.
Arm/Group | Satiators | Sensitizers
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/36
Other Adverse Events (participants affected / at risk) | 0/165 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT04027608/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT04027608/SAP_001.pdf
  • Informed Consent Form (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT04027608/ICF_002.pdf